CLINICAL TRIAL: NCT02612636
Title: The Effect of Ear Plug and Eye Mask on Sleeping Quality in Critically Ill Patients
Acronym: sayed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Professor (Anesthesiology and Critical Care)- College of Medicine-Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB0000871100
Record Dates: First submitted 2015-11-16; First posted 2015-11-24 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Sleep
Keywords: Delirium; Ear Plug; Eye Mask; Mechanical ventilation; Sleep
MeSH Terms: conditions — Delirium | interventions — Ear Protective Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ear plug and eye mask (Active Comparator): * The patients will not receive the intervention in the first night (N1) from 9 pm to 6 am
  * The patients will receive the intervention (eye mask) in the second night (N2) from 9 pm to 6 am.
  * The patients will receive the intervention (ear plug) in the third night (N3) from 9 pm to 6 am.
  * The patients will receive the intervention (eye mask and ear plug) in the fourth night (N4) from 9 pm to 6 am.
  Interventions: Other: ear plug; Other: eye mask
- control (No Intervention): The researcher will assess and observe the patients who are receiving the routine hospital nursing care during the four nights.

INTERVENTIONS:
Other: ear plug — The patients will receive the intervention (ear plug) in the third night (N3) from 9 pm to 6 am.
  Other Names: eastnova ear plug
  Arms: ear plug and eye mask
Other: eye mask — The patients will receive the intervention (eye mask) in the second night (N2) from 9 pm to 6 am.
  Other Names: Sleeping mask
  Arms: ear plug and eye mask

SUMMARY:
Sleep is a complex physiologic and behavioral process essential for rest, repair, well-being, and survival. Sleep is defined as a periodic, reversible state of cognitive and sensory disengagement from the external environment. Critically ill patients experience poor sleep quality. Surveys of ICU survivors have shown that sleep disruption, pain and intubation for mechanical ventilation are the major sources of anxiety and stress during the ICU stay. Many physiological, psychological and environmental factors contribute to the incidence of sleep disruption for the ICU patients. The primary physiologic factors documented in the literature are pain, medications and illness.The primary psychological factors documented in the literature are stress and worry. Environmental factors include noise, patient care activities and therapeutic modalities as mechanical ventilation. Our research aim will be the impact of effective interventions like use of ear plugs and eye mask on decreasing light exposure and promoting sleep in ICU patients.

DETAILED DESCRIPTION:
50 patients in the age range 18- 60 years admitted to ICU of Assiut university hospitals will be randomly allocated into into two groups (control group and intervention group).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old.
* Mechanically ventilated patient.
* Conscious patient.
* No hearing problems.
* No eye disease.
* Not receiving narcotic drugs five to six hours before sleep time at night.
* No underlying disease that is affecting sleep such as rheumatoid arthritis and migraine.

Exclusion Criteria

* Head injury.
* Psychiatric disease.
* Shocked patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Sleep quality . | four days
  to assess sleep quality by using quality of sleep questionnaire or the Richards-Campbell Sleep Questionnaire (RCSQ) (measured by Units on a Scale)

SECONDARY OUTCOMES:
Urine Melatonin | four days
  as urine Melatonin ( pg/mL)
Cortisol level | four days
  stress hormone as cortisol level (nmol/L)
Delirium assessment | four days
  Assessment of delirium by using NEECHAM confusion scale or Nursing delirium screening scale (measured by Units on a Scale)

CONTACTS AND LOCATIONS:
Overall Officials: sayed abd elshafy, Principal Investigator — associate professor
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided